CLINICAL TRIAL: NCT07216820
Title: Interscalene vs Phrenic-sparing Blocks in Obesity: Effect of Pre-operative Maximum Inspiratory Pressure in a Randomized Trial
Brief Title: Interscalene vs Phrenic-sparing Blocks in Obesity and Effect of Maximum Inspiratory Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Society of Regional Anesthesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-3332
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Surgery; Obesity
Keywords: interscalene block; phrenic-sparing block; brachial plexus block
MeSH Terms: conditions — Obesity | interventions — Bupivacaine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Standard Interscalene Block (Active Comparator): Standard Interscalene Brachial Plexus Block (Control)
  Description:
  Participants receive a single 16 mL interscalene block at the C5-C6 level under ultrasound guidance. The injectate contains 15 mL of 0.5% bupivacaine HCl (75 mg) mixed with 1 mL preservative-free dexamethasone (4 mg).
  Interventions: Procedure: Ultrasound-Guided Interscalene Brachial Plexus Block; Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Dexamethasone 4mg
- Arm 2: Phrenic-Sparing Block Combination (Experimental): Combined Infraclavicular + Distal Suprascapular Block (Phrenic-Sparing Technique)
  Description:
  Participants receive two ultrasound-guided peripheral nerve blocks designed to minimize phrenic nerve involvement:
  Infraclavicular block: 15 mL 0.5% bupivacaine + 1 mL dexamethasone (total 16 mL) Distal suprascapular block: 12 mL 0.5% bupivacaine + 1 mL dexamethasone (total 13 mL) Total local-anesthetic dose = 135 mg bupivacaine + 8 mg dexamethasone, within accepted safety limits.
  Interventions: Procedure: Phrenic-Sparing Block Combination (Experimental); Drug: Bupivacaine HCl 0.5% Injectable Solution; Drug: Dexamethasone 4mg

INTERVENTIONS:
Procedure: Ultrasound-Guided Interscalene Brachial Plexus Block — Single 16 mL injection (15 mL 0.5 % bupivacaine + 1 mL dexamethasone 4 mg) at the C5-C6 root level under ultrasound guidance.
  Performed pre-operatively as standard care for shoulder surgery. Arm Cross-Reference: Standard Interscalene Block (Control)
  Arms: Arm 1: Standard Interscalene Block
Procedure: Phrenic-Sparing Block Combination (Experimental) — Infraclavicular: 15 mL (75 mg) 0.5 % bupivacaine + 1 mL dexamethasone (4 mg) injected around the cords of the brachial plexus beneath the clavicle under ultrasound guidance.
  Distal Suprascapular: 12 mL (60 mg) 0.5 % bupivacaine + 1 mL (4 mg) dexamethasone injected at the suprascapular notch under ultrasound guidance to provide complete shoulder coverage while minimizing phrenic nerve involvement. Total local anesthetic dose = 135 mg bupivacaine + 8 mg dexamethasone.
  Arm Cross-Reference: Phrenic-Sparing Block Combination (Experimental)
  Arms: Arm 2: Phrenic-Sparing Block Combination
Drug: Bupivacaine HCl 0.5% Injectable Solution — Infraclavicular: Adminstered as 15 mL (75 mg) injection (together with dexamethasone).
  Distal Suprascapular: Adminstered as 12 mL (60 mg) injection (together with dexamethasone).
  Other Names: Bupivacaine Hydrochloride Injection
Drug: Dexamethasone 4mg — Adminstered as applicable for infraclavicular and distal suprascapular: as 1 mL (4 mg) injection (together with bupicacaine 0.5%).
  Other Names: Decadron, Dexamethasone Intensol, De-Sone LA, Dxevo, Dexacorten

SUMMARY:
The goal of this clinical trial is to learn whether a phrenic-sparing nerve block can lower early breathing problems after shoulder surgery in adults with obesity, and whether a simple breathing-strength test (maximum inspiratory pressure, MIP) helps identify who is at higher risk. The main questions are:

Does the phrenic-sparing approach reduce breathlessness or oxygen need in the recovery room (30-60 minutes after arrival)? Do patients have similar pain control and opioid use compared with the standard interscalene block (ISB)? Are there any breathing-related complications or unplanned admissions within 24 hours? Researchers will compare the phrenic-sparing block (infraclavicular + distal suprascapular) to the standard ISB, both commonly used at UNC.

Participants will:

Have a quick MIP breath test before surgery (and, if age ≥65, a brief thigh muscle ultrasound).

Be randomly assigned to receive either the standard ISB or the phrenic-sparing block (both ultrasound-guided and part of routine care).

Receive usual anesthesia/surgery; have a brief recovery check at 30-60 minutes (breathlessness score, oxygen use, oxygen level).

Have pain medicines recorded from anesthesia start to PACU discharge; the team may review the chart up to 24 hours and make a short follow-up call (24-48 hours).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (self-report, confirmed on chart).
* Body-mass index ≥ 35 kg m^2 at the pre-operative clinic visit (chart).
* Scheduled for elective unilateral shoulder surgery (arthroscopy, arthroplasty, rotator cuff repair, reverse arthroplasty) under general anesthesia at UNC Hospitals
* Planned use of a single-injection regional brachial-plexus block for postoperative analgesia (anesthesia record).
* Able to perform a maximal-inspiratory-pressure (MIP) maneuver at screening, producing two reproducible efforts (bedside test)
* Able to read or understand English and provide written informed consent (consent discussion).

Exclusion Criteria:

* Emergent or trauma shoulder procedure or case converted to open surgery (schedule/chart).
* Pregnancy confirmed by point-of-care urine test on day of surgery (POC test). Prisoner status or legal incapacity to consent (chart/interview).
* Severe pulmonary disease: GOLD stage 3-4 COPD, restrictive lung disease unrelated to obesity with FVC < 50 % predicted, baseline dyspnea Borg ≥ 3, or home oxygen therapy (pulmonary clinic notes, patient interview).
* Severe heart disease- Severe valvular heart disease, Congestive Heart Failure NYHA Class III or IV, Obstructive Coronary Artery Disease with Angina
* Neuromuscular disorders affecting respiratory muscles (e.g., ALS, myasthenia gravis) or known diaphragmatic paralysis (chart).
* Coagulopathy (platelets < 100 × 10/ L or INR > 1.5) or local infection at block sites (pre-op labs/assessment).
* Anemia and hemoglobinopathies: Hgb <10 g/dl, clinically significant hemoglobinopathy.
* Allergy to bupivacaine, dexamethasone, or ultrasound gel (self-report).
* Chronic opioid use > 100 mg oral-morphine equivalents per day in the three months preceding surgery (medication history, PDMP query).
* Prior enrolment in this trial or planned participation in another interventional study that might confound outcomes (research registry).
* Anticipated inability to comply with postoperative assessments (e.g., profound cognitive impairment, expected early transfer to outside facility) as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Early Postoperative Respiratory Compromise | Within 60 minutes after arrival to PACU
  Composite outcome defined as either (a) a Modified Borg Dyspnea Score ≥ 3 in the post-anesthesia care unit (PACU, 30-60 minutes after surgery) or (b) continued need for supplemental oxygen at the PACU assessment.
  Outcome Type: Primary Unit of Measure: Percentage of participants meeting composite endpoint.
Effect Modification by Preoperative Maximum Inspiratory Pressure (MIP) | Baseline (preoperative MIP test) and PACU assessment (30-60 minutes post-surgery).
  Assess whether the magnitude of treatment benefit from the phrenic-sparing block varies by baseline inspiratory-muscle strength. The effect is modeled as the interaction between block type and continuous MIP (cm H₂O) on the composite respiratory-compromise endpoint.
  Unit of Measure: Interaction odds ratio (per 10 cm H₂O decrement in MIP).

SECONDARY OUTCOMES:
Lowest Oxygen Saturation (SpO₂) in PACU | From PACU arrival to discharge (typically 60-120 minutes)
  Minimum oxygen saturation recorded by pulse oximetry during the PACU stay Unit of Measure: Percent (%)
Total Duration of Supplemental Oxygen Use | 0-24 hours post-surgery.
  Total number of hours on oxygen from PACU arrival until hospital discharge (maximum 24 hours).
  Unit of Measure: Hours.
Post-Induction Opioid Consumption | 0-6 hours post-surgery.
  Total opioid dose administered from anesthesia induction to PACU discharge, converted to oral morphine milligram equivalents (OMME).
  Unit of Measure: mg OMME.
Diaphragmatic Excursion Change from Baseline | Baseline (pre-block) and 30-60 minutes post-surgery in PACU.
  Percent change in diaphragmatic excursion (ultrasound-measured) from baseline to PACU.
  Unit of Measure: Percent change (%).
PACU Pain Score | Within 1 hour after PACU arrival.
  Numeric Rating Scale (NRS) for pain recorded at 30-60 minutes post-surgery. Unit of Measure: 0-10 NRS scale.

OTHER OUTCOMES:
Exploratory: Association of Frailty and Sarcopenia Measures With Respiratory Outcomes | Baseline preoperative assessment; outcome analyzed at PACU.
  Explore whether rectus femoris index (cm/height²) or Clinical Frailty Scale (CFS) scores predict postoperative respiratory compromise in participants ≥ 65 years.
  Unit of Measure: Correlation coefficient or adjusted risk ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Nanda, Principal Investigator — University of North Carollina at Chapel Hill
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.